CLINICAL TRIAL: NCT00910871
Title: A Phase II, Open-label Trial With TMC207 as Part of a Multi-drug Resistant Tuberculosis (MDR-TB) Treatment Regimen in Subjects With Sputum Smear-positive Pulmonary Infection With MDR-TB.
Brief Title: To Evaluate the Safety, Tolerability, and Efficacy of TMC207 as Part of an Individualized Multi-drug Resistant Tuberculosis (MDR-TB) Treatment Regimen in Participants With Sputum Smear-positive Pulmonary MDR-TB.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012352; TMC207-TiDP13-C209 (Other: Janssen Infectious Diseases BVBA); 2008-008444-25 (EudraCT Number); NCT00980811 (obsolete NCT alias)
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TMC207-TiDP13-C209; TMC207-C209; TMC207; TB; MDR-TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMC207 (Experimental): TMC207 400mg once daily for 2 weeks then 200mg three times a week for 22 weeks in addition to Background Regimen (BR) for the treatment of multi-drug resistant tuberculosis (MDR-TB).
  Interventions: Drug: TMC207; Drug: Background Regimen (BR) for MDR-TB

INTERVENTIONS:
Drug: TMC207 — TMC207 400mg once daily for 2 weeks then 200mg three times a week for 22 weeks.
Drug: Background Regimen (BR) for MDR-TB — Background Regimen (BR) of antibacterial drugs used in the treatment of TB according to national TB program and selected at the baseline visit as specified in the protocol for up to 96 weeks.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of TMC207 in combination with an individualized background regimen (BR) of antibacterial drugs as treatment for MDR-TB

DETAILED DESCRIPTION:
This is a Phase II, open-label (all people involved know the identity of the intervention) trial to evaluate the safety, tolerability, and efficacy of TMC207 as part of an individualized Multi-drug Resistant Tuberculosis (MDR-TB) treatment regimen in participants with sputum smear-positive pulmonary MDR-TB. Approximately 225 participants will receive TMC207 for 24 weeks in combination with an individualized background regimen (BR) of antibacterial drugs used in the treatment of TB according to national and international guidelines and selected at the baseline visit. TMC207 dosage will be 400 mg once daily (q.d.) for the first 2 weeks and 200 mg 3 times/week (t.i.w.) for the following 22 weeks. Upon completion of the 24-week treatment with TMC207, all participants will continue to receive their BR under the care of their physician and in accordance with national TB program (NTP) treatment guidelines.

Additionally, the pharmacokinetics (how the body absorbs, distributes, metabolizes and eliminates a drug) of TMC207 and its N-monodesmethyl metabolite (M2), and pharmacokinetic/pharmacodynamic (the study of the action or effects a drug has on the body) relationships for safety and efficacy will be assessed. Safety evaluations that will be performed are lab tests, vital signs, ECG, reporting of adverse events, physical examinations and X-rays.

All participants will be followed up for 19 months after their last intake of TMC207. Also participants who prematurely withdraw (unless they withdraw consent) will be followed for this period or until the last follow-up visit for the last patient in the trial. Investigators will be asked to provide information about the survival/clinical outcome of these participants throughout the follow-up period, approximately every 6 months.

Primary outcome is time to sputum culture conversion in Mycobacteria Growth Indicator Tube (MGIT) during and beyond treatment with TMC207. Sputum culture conversion will be defined as 2 consecutive negative cultures from sputa collected at least 28 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Females of child-bearing potential must be using and are willing to continue using effective birth control methods, or be willing to practice sexual abstinence throughout treatment or be nonheterosexual active
* Confirmed pulmonary MDR-TB infection including those infected with XDR (extensively drug resistant)-TB
* Positive for acid-fast bacilli (AFB) on direct smear examination of expectorated sputum specimen (= 1+ smear-positive)
* HIV-positive patients are eligible, provided they meet the requirements as described in the protocol
* Must voluntarily sign the Informed Consent Form (ICF) prior to starting any study activities
* Willing to comply with protocol requirements
* Willing to comply with NTP treatment guidelines

Exclusion Criteria:

* Patients having a known or suspected hypersensitivity or serious adverse reaction to TMC207
* Patients with significant cardiac arrhythmia requiring medication
* Patients with complicated or severe extrapulmonary manifestations of TB, including central nervous system infection
* Patients with certain QT/QTc interval characteristics as described in the protocol
* Patients having participated in other clinical studies with investigational agents, within 8 weeks prior to trial start
* Women who are pregnant or breastfeeding
* Patients who have previously received treatment with TMC207 as part of a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (27):
- China (5):
  - Beijing
  - Fuzhou
  - Jinan
  - Nanjing
  - Shanghai
- Estonia (2):
  - Talinn
  - Tartu
- Nairobi, Kenya
- Stopinu Region, Latvia
- Peru (2):
  - Callao
  - Lima
- Quezon City, Philippines
- Russia (3):
  - Arkhangelsk
  - Moscow
  - Oryol
- South Africa (3):
  - Bellville West Cape
  - Durban
  - Sandringham
- South Korea (2):
  - Seoul
  - Suwon
- Thailand (2):
  - Nakhon
  - Nonthaburi
- Turkey (Türkiye) (2):
  - Istanbul
  - Keçiören
- Ukraine (3):
  - Donetsk
  - Kiev
  - Odesa

REFERENCES:
- [Derived] Bolhuis MS, Akkerman OW, Sturkenboom MGG, van Boven JFM, Alffenaar JC, Stevens J. Bedaquiline exposure in people with drug-resistant TB treated for diabetes: analysis of two phase 2 trials. Int J Tuberc Lung Dis. 2023 Apr 1;27(4):335-337. doi: 10.5588/ijtld.22.0581. No abstract available. PMID 37035978
- [Derived] Pym AS, Diacon AH, Tang SJ, Conradie F, Danilovits M, Chuchottaworn C, Vasilyeva I, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, Van Baelen B, van Heeswijk RP, Dannemann B; TMC207-C209 Study Group. Bedaquiline in the treatment of multidrug- and extensively drug-resistant tuberculosis. Eur Respir J. 2016 Feb;47(2):564-74. doi: 10.1183/13993003.00724-2015. Epub 2015 Dec 2. PMID 26647431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase II open label trial with TMC207 as part of multi-drug resistant mycobacterium tuberculosis (MDR-TB) treatment regimen in participants with sputum smear-positive pulmonary infection with MDR-TB.
Pre-assignment Details: A total of 241 participants were enrolled in the study; 8 participants were withdrawn from the study before study drug administration and 233 started treatment with study drug.
Groups:
- TMC207: Participants will receive 400 milligram (mg) TMC207 tablets orally 2 times a day along with background regimen from Day 1 to Week 2 followed by 200 mg TMC207 tablets orally 3 times a day from Week 3 to Week 24 along with background regimen, then background therapy from Week 25 to end of study (Week 120).
Period: Overall Study
Arm/Group | TMC207
Started | 233
Completed | 179
Not Completed | 54
Not completed — Adverse Event | 5
Not completed — Death | 12
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 12
Not completed — Subject didn't meet eligibility criteria | 5
Not completed — Undefined | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who had at least 1 dose of TMC207, regardless of their compliance with the protocol.
Arm/Group | TMC207
Number analyzed (Participants) | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 150

OUTCOME MEASURES:

1. Primary Outcome: The Median Time to Sputum Culture Conversion
Description: The table below shows the median time in days to culture conversion for the modified intent-to-treat (mITT) population up to Week 24. Sputum culture conversion is defined as 2 consecutive sputum cultures negative for multi-drug resistant tuberculosis (MDR-TB) taken at least 25 days apart. Participants who discontinued during the 24-week period were considered non-responders (based on Mycobacteria Growth Indicator Tube [MGIT]).
Time Frame: Up to Week 24
Population: The modified intent-to-treat (mITT) population used for all efficacy analyses included all randomized participants who received at least 1 dose of TMC207 excluding participants with drug-susceptible tuberculosis (DS-TB) or participants that were not evaluable for efficacy.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC207
Number analyzed (Participants) | 205
Days | 57 [56.00 to 83.00]

2. Secondary Outcome: The Percentage of Participants With Sputum Culture Conversion
Description: The table below shows the percentage of participants who were responders to treatment. Sputum culture conversion is defined as 2 consecutive sputum cultures negative for multi-drug resistant tuberculosis (MDR-TB) taken at least 25 days apart. Participants who discontinued or died during the trial were considered non-responders.
Time Frame: Week 120
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC207
Number analyzed (Participants) | 205
Percentage of Participants | 72.2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 120
Description: Only participants who had at least one of the treatment emergent adverse events (TEAEs) listed in the other (non-serious) adverse events table are included in the total number of participants with non-serious adverse events.
Arm/Group | TMC207
Serious Adverse Events (participants affected / at risk) | 47/233
Other Adverse Events (participants affected / at risk) | 179/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207 (N=233)
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Cor pulmonale (Cardiac disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Treatment failure (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Tuberculosis (Infections and infestations) | 6
Blood glucose fluctuation (Investigations) | 1
Electrocardiogram qt prolonged (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Emotional disorder (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Surgery (Surgical and medical procedures) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatitis a (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lymph node tuberculosis (Infections and infestations) | 1
Pyopneumothorax (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Lung operation (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207 (N=233)
Tinnitus (Ear and labyrinth disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 26
Injection site pain (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 17
Blood uric acid increased (Investigations) | 20
Hyperuricaemia (Metabolism and nutrition disorders) | 36
Hypokalaemia (Metabolism and nutrition disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 35
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 31
Insomnia (Psychiatric disorders) | 18
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 18
Anaemia (Blood and lymphatic system disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 14
Chest pain (General disorders) | 17
Upper respiratory tract infection (Infections and infestations) | 13
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 14
Hepatic enzyme increased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Rash (Skin and subcutaneous tissue disorders) | 13

LIMITATIONS AND CAVEATS:
In Participant Flow, the 12 deaths shown are restricted to those that occurred during the trial and do not include 4 deaths reported after discontinuation in long-term survival follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is the policy of the sponsor not to allow the investigators to publish their results or findings prior to the sponsor's publication of the overall trial results.The investigator agrees that before he/she publishes any results of this trial, he/she shall provide the sponsor with at least 45 days for full review of the prepublication manuscript prior to submission of the manuscript to the publisher.